CLINICAL TRIAL: NCT00726635
Title: Assessment of the Impact of Preoperative Stress Reduction on Psychological, Physiological and Immunological Parameters in Women With Gynecological Malignancies - Prospective Randomized Controlled Trial
Brief Title: The Assessment of Preoperative Psychological Intervention on Stress in Women With Gynecological Malignancies
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Academic College of Tel Aviv-Jaffa (Other); Israel Cancer Association (Other)
Responsible Party: Opher Caspi, MD PhD, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0014-08-RMC
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Last update posted 2009-02-17 (Estimated); Status verified 2008-07

CONDITIONS: Cancer of Cervix; Ovarian Cancer; Cancer of Endometrium
MeSH Terms: conditions — Uterine Cervical Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Women in this arm will not receive a psychological intervention but rather will have a conversation with a nurse for one hour (attention control).
  Interventions: Other: Control group
- 2 (Experimental): Cognitive intervention: Women in this arm will receive a cognitive psychological intervention(cognitive technique:self-talk)
  Interventions: Behavioral: Cognitive intervention
- 3 (Experimental): Psycho-physiological intervention: Women in this arm will receive a psycho-physiological intervention (relaxation and guided imagery)
  Interventions: Other: psycho-physiological intervention

INTERVENTIONS:
Behavioral: Cognitive intervention — The intervention will last one hour and will include cognitive technique (self-talk). The technique will be demonstrated to the woman, practiced with her, and taped so as to encourage further practice at home.
  Other Names: Tailored cognitive intervention
  Arms: 2
Other: Control group — A one hour conversation with a nurse
  Arms: 1
Other: psycho-physiological intervention — The intervention will last an hour and will include a psycho-physiological intervention (relaxation and guided imagery). The technique will be demonstrated to the woman, practiced with her, and taped so as to assure further practice at home
  Other Names: tailored psycho-physiological intervention
  Arms: 3

SUMMARY:
The purpose of this study is to asses the impact of a tailored preoperative psychological intervention on women with gynecological malignancies on psychological, physiological and immunological parameters

DETAILED DESCRIPTION:
Surgery is considered one of the most stressful events in human life. Research indicates that patients show high levels of stress from at least six days before surgery and up to a week post the operation. Stress levels return to normalcy only after several weeks. Research shows that psychological interventions given to women suffering from cancer can improve their coping abilities and overall function, decreases stress levels, enhances adherence to treatments,and increases quality of life and even life expectancy.

Women enrolled in this study will be divided into two groups: an experimental group and a control group. Both groups will receive standard care. The control group will interact with a nurse for one hour. The experimental group will receive one of two forms of psychological intervention: either a cognitive intervention, or a psychophysiological intervention (tailored to each woman).

Measurements and Instruments include: 1) Self-report questionnaires, such as:Profile of Mood States (POMS-SF),Coping Inventory (COPE), Life Orientation Test Revised (LOT- R),Stress Level Report, 2) Demographics, 3) Global assessment by the head nurse. 4)Physiological and behavioral measures, such as: vital signs and use of medicine. 5)Hormonal and immunological measures: levels of cortisol in saliva and plasma, levels of catecholamines in plasma, salivary levels of IgA1, and peripheral blood NK cells and lymphocyte phenotyping.6)levels of cytokines including IL-1,2,4,6,10,12, TNF-alpha, Interferon-gamma.

Time intervals for the collection of blood and saliva and the administration of the questionnaires:

During the first week after being given the diagnosis and prior to the intervention:Blood & saliva, Stress Level Report, POMS-SF, COPE, LOT-R

A day prior to surgery:Blood & saliva, Stress Level Report

On discharge from hospital:Blood & saliva, Stress Level Report

30 days after surgery:Stress Level Report,POMS-SF,COPE,LOT-R.

ELIGIBILITY:
Inclusion Criteria:

* Woman with ovarian, cervical or endometrial cancer/tumor
* Women who speak Hebrew
* Women who sign the consent form

Exclusion Criteria:

* Women who have received neoadjuvant treatment
* Women suffering from any form of depression, anxiety or schizophrenia
* Women suffering from autoimmune or infectious diseases
* Women taking medications which have immunological effects (steroids ,beta-blockers)
* Women suffering from dementia or concentration problems

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-08 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
psychological, physiological, immunological parameters | A week before surgery, the day befor surgery, day of hospital discharge, one month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Opher Caspi, MD PhD, Principal Investigator — Director, Integrative Medicine - Rabin Medical Center
Locations (1):
- Rabin Medical center, Petah Tikva, Israel